CLINICAL TRIAL: NCT00883857
Title: Comparison Endotracheal Cardiac Output Monitor (ECOM) to a Standard Device in Measuring Heart Blood Volume
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Aman Mahajan, Principal Investigator, University of California, Los Angeles
Other Study IDs: 06-04-090-03
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Heart Disease; Cardiac Surgery
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate a new monitor that measures cardiac output (amount of blood pumped by the heart). The system that is being tested in this study, called Endotracheal Cardiac Output Monitor (ECOM), uses electricity (impedance cardiography) to measure cardiac output and is not harmful to the patient.

This study will test the accuracy and efficacy of the ECOM system in anesthetized and sedated patients who, in the normal course of clinical care in the OR or ICU, are having cardiac output measured. The investigators propose that unlike the standard system for cardiac output measurement, the ConMed ECOM System should result in a simplified, inexpensive, continuous, less-invasive, and accurate method of measuring cardiac output. Such a technique could allow the rapid diagnosis of instability in the cardiovascular system for critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Patients requiring all of the following:

  * an oral ET tube
  * an arterial catheter
  * measurement of CO

Exclusion Criteria:

* Patients not competent to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for cardiac surgery
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aman Mahajan, MD, PhD, Study Director — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States